CLINICAL TRIAL: NCT05077878
Title: Dentine Sialophosphoprotein (DSPP) Quantification for Root Resorption Prediction Using Multivariate Versus Univariate Spectrum Analysis
Brief Title: Analysis of Dentine Sialophosphoprotein (DSPP) for Root Resorption
Status: Completed | Type: Observational
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Rohaya Megat Abdul Wahab, Professor, National University of Malaysia
Other Study IDs: UKMfggRMAW
Record Dates: First submitted 2021-09-30; First posted 2021-10-14 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Root Resorption
Keywords: DSPP
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normal: Patients with non-orthodontic treatment and have no root resorption
  Interventions: Biological: DSPP level in GCF
- mild to moderate: Patients with orthodontic treatment and have mild to moderate root resorption
  Interventions: Biological: DSPP level in GCF
- severe: Child patients with non-orthodontic treatment and have severe root resorption
  Interventions: Biological: DSPP level in GCF

INTERVENTIONS:
Biological: DSPP level in GCF — quantification of DSPP
  Other Names: Root resorption

SUMMARY:
This study was conducted after obtaining approval from UKM Research Ethics Committee. Gingival Crevicular Fluid (GCF) from Orthodontic and non-orthodontic patients was collected with the consent of patients to detect Dentine sialophosphoprotein. Spectrometry analysis of Gingival Crevicular Fluid was conducted in collaboration with MIMOS Berhad.

DETAILED DESCRIPTION:
Thirty patients were recruited having met the following inclusion criteria of (1) good general health, (2) good periodontal health, (3) caries-free, (4) good oral hygiene. The subjects were divided into 3 groups based on a radiographic assessment on the level of root resorption; normal (no root resorption), mild (less than 2 mm), and severe (more than 2 mm). The GCF samples were taken from the permanent central incisors of untreated subjects in the normal control group (n=14), while in the mild group, samples were collected from the permanent central incisors with mild root resorption (<2 mm) in patients undergoing active orthodontic treatment after 6 months with radiographic evidence (mild group, n=5). Child patients with severe root resorption (>2 mm) were those with primary second molars undergoing physiological root resorption (severe group, n=11). The GCF samples were collected from the mesial and the distal gingival crevicular sulcus of the involved teeth using gingival fluid collection strips (Periopaper, Oraflow, Smithtown, N.Y.). The paper strips were placed within the sulcus (intrasulcular method) approximately 1 to 2 mm into the gingival sulcus and left in situ for 60 seconds. Every sample collection was taken 3 times at the same site with one-minute resting intervals to allow GCF to be replenished into the gingival sulcus.

ELIGIBILITY:
Inclusion Criteria:

* good general health,
* good periodontal health,
* caries-free,
* good oral hygiene

Exclusion Criteria:

* Consumption of anti-inflammatory drugs and antibiotics

Ages: 10 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients that come to the dental clinic for treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
value of wavelength of DSPP in GCF from non-orthodontic patient with no root resorption | 1 month
  The absorbance values at a single wavelength at 450 nm
value of wavelength of DSPP in GCF from orthodontic patient with mild to moderate root resorption | 1 month
  The absorbance values at a single wavelength at 450 nm
value of wavelength of DSPP in GCF from child patient severe root resorption | 1 month
  The absorbance values at a single wavelength at 450 nm

CONTACTS AND LOCATIONS:
Overall Officials: Rohaya Megat Abdul Wahab, Master, Principal Investigator — Faculty of Dentistry, Universiti Kebangsaan Malaysia
Locations (1):
- Faculty of Dentistry, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mohd Zain MN, Md Yusof Z, Basri KN, Yazid F, Teh YX, Ashari A, Zainal Ariffin SH, Megat Abdul Wahab R. Multivariate versus univariate spectrum analysis of dentine sialophosphoprotein (DSPP) for root resorption prediction: a clinical trial. BMC Oral Health. 2022 Apr 29;22(1):151. doi: 10.1186/s12903-022-02178-2. PMID 35488332